CLINICAL TRIAL: NCT05965596
Title: Effect of a Psycho-educational Intervention on Psychological Outcomes and Quality of Life Among Gynecological Cancer Patients in El-shatby University Hospital, Alexandria: Randomized Controlled Trial
Brief Title: Effect of a Psycho-educational Intervention on Psychological Outcomes of Gynecological Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: psycho-educational
Record Dates: First submitted 2023-07-11; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Psychological
Keywords: gynecological cancer; quality of life

STUDY DESIGN:
Intervention Model Description: a randomly selected sample of gynecological cancer women attending the study setting, fulfilling the inclusion criteria and consented to participate in the study will be recruited into the study sample. Then they will be randomly assigned into either the intervention group or the control group using computer-generated random codes in serially numbered opaque sealed envelopes. Creation and concealment of the allocation sequence will be done by the supervisor. While the researcher will enroll the participants, assess eligibility, discuss the trial, obtain consent, ascertain intervention assignment (such as opening next envelope) and carry out the intervention. Participants in the intervention group will receive a psycho educational intervention program and those in the control group will receive the routine care provided for all gynecological cancer patients in the study setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Experimental): Participants in the intervention group will receive a psychoeducational intervention program
  Interventions: Other: a psycho educational intervention program
- the control group (Sham Comparator): those in the control group will receive the routine care provided for all gynecological cancer patients in the study setting.
  Interventions: Other: the routine care

INTERVENTIONS:
Other: a psycho educational intervention program — The program was developed by the researcher herself based on recommendations derived from a systematic review of psychoeducational interventions to improve the quality of Life and psychological outcomes in gynecological cancer patients. Also guided by the program adopted by chow et all in 2014(28) to test the feasibility of implementing a psychoeducational intervention program for gynecological cancer patients.
  Arms: the intervention group
Other: the routine care — the routine care provided for all gynecological cancer patients in the study setting
  Arms: the control group

SUMMARY:
This study will be conducted to optimize the quality of care rendered for gynecological cancer patients attending the Gynecological Oncology Unit in El-Shatby University Hospital in Alexandria.As well as to assess the effect of implementing a psychoeducational intervention program among gynecological cancer women on the:

1. Quality of life with its different domains (physical, emotional, social and functional). "as a primary objective"
2. Psychological distress and cancer-specific stress. "as secondary objectives"

DETAILED DESCRIPTION:
Cancer is a significant health problem worldwide with wide geographical variation in incidence. Additionally it has become an important item in each country's health agenda.It is a prominent cause of mortality in both economically developed and underdeveloped nations.Unfortunately, the burden is expected to grow globally due to the development and aging of the population.Gynecological cancer, which includes cancers of the cervix, ovary, uterus, vulva, vagina and fallopian tube are among the leading causes of cancer-related mortality worldwide.In Egypt, according to the Global Cancer Observatory (GLOBOCAN) 2020, approximately 2,787 new cases for ovarian cancer were diagnosed and 1,839 women died from the disease,1,694 new cases for uterine cancer and 350 women died from the disease and 1,320 new cases for cervical cancer and 744 women died from the disease.

Hence, this study will be carried out to develop and implement a psychoeducational intervention program among gynecological cancer patients attending the Gynecological Oncology Unit in El-Shatby University Hospital in Alexandria and evaluate its effect in improving their psychological outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Women are eligible to participate if they are:

* Over 20 years old.
* Newly diagnosed cases with gynecological cancers (confirmed within 3 months).
* Scheduled to have surgery as the first-line treatment.
* Willing to participate in the study.

Exclusion Criteria:

Women are excluded if they:

* Are in the late stage (stage IV) as women in this group usually receive palliative/ symptomatic treatment.
* Have additional cancer diagnosis (including metastasis).
* Are diagnosed with severe psychiatric or cognitive disorder.
* Participate in other intervention study.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
A change in the Quality of life of gynecological cancer patients | over approximately 2 months for each patient as the tool is used initially before surgery and reused 8 weeks after the operation
  A change in the Quality of life from baseline and follow up sessions is assessed using the Arabic version of the Functional Assessment of Cancer Therapy-General (FACT-G) version 4. It includes 27 items and covers four primary QOL domains: physical wellbeing (PWB; 7 items, score range 0-28), emotional well-being (EWB; 6 items, score range 0-24), social well-being (SWB; 7 items, score range 0-28) and functional well-being (FWB; 7 items, score range 0-28). A five-point Likert scale will be used (0 = not at all, 1 = a little bit, 2 = somewhat, 3 = quite a bit, 4 = very much), which provided four subscale scores and a total score ranging from 0 to 108, a higher score meaning a poor QOL, a lower score indicating high QOL and low effect of gynecological cancer treatment on QOL.

SECONDARY OUTCOMES:
A change in the Anxiety and depression | over approximately 2 months for each patient as the tool is used initially before surgery and reused 8 weeks after the operation
  A change in the psychological distress from baseline and follow up sessions is assessed using the Arabic version of the Hospital Anxiety and Depression Scale (HADS).There is a total of 14 items in the scale which are equally distributed into anxiety and depression subscales. Higher scores reflect greater psychological distress.
A change in the Cancer-specific stress | over approximately 2 months for each patient as the tool is used initially before surgery and reused 8 weeks after the operation
  A change in the traumatic stress reactions to cancer diagnosis and treatment from baseline and follow up sessions is assessed using The Impact of Events Scale-Revised (ӀEЅ-R).The participants will be asked to rate the frequency of these feelings or events during the previous week, using а five-point Likert scale ranging from 0 = not at all to 4 = extremely. Items will be summed for а total score that ranges from 0 to 88. The IES-R is not meant to be diagnostic. While there is no specific cut-off score, scores higher than 24 are of concern; the higher the score the greater the concern for PTSD and associated health and well-being consequences.

CONTACTS AND LOCATIONS:
Overall Officials: faculty of medicine Alexandria university, Study Director — Alexandria University
Locations (1):
- El-Shatby University Hospital, Alexandria, Bab Sharqi, Egypt

REFERENCES:
- [Background] Chow KM, Chan JC, Choi KK, Chan CW. A Review of Psychoeducational Interventions to Improve Sexual Functioning, Quality of Life, and Psychological Outcomes in Gynecological Cancer Patients. Cancer Nurs. 2016 Jan-Feb;39(1):20-31. doi: 10.1097/NCC.0000000000000234. PMID 25730595
- [Background] Tangjitgamol S, Manusirivithaya S, Hanprasertpong J, Kasemsarn P, Soonthornthum T, Leelahakorn S, Thawaramara T, Lapcharoen O. Sexual dysfunction in Thai women with early-stage cervical cancer after radical hysterectomy. Int J Gynecol Cancer. 2007 Sep-Oct;17(5):1104-12. doi: 10.1111/j.1525-1438.2007.00907.x. Epub 2007 Mar 15. PMID 17367316
- [Background] Padilla GV, Ferrell B, Grant MM, Rhiner M. Defining the content domain of quality of life for cancer patients with pain. Cancer Nurs. 1990 Apr;13(2):108-15. PMID 2331691
- [Background] Lim JW, Yi J, Zebrack B. Acculturation, social support, and quality of life for Korean immigrant breast and gynecological cancer survivors. Ethn Health. 2008 Jun;13(3):243-60. doi: 10.1080/13557850802009488. PMID 18568975
- [Background] Weaver KE, Forsythe LP, Reeve BB, Alfano CM, Rodriguez JL, Sabatino SA, Hawkins NA, Rowland JH. Mental and physical health-related quality of life among U.S. cancer survivors: population estimates from the 2010 National Health Interview Survey. Cancer Epidemiol Biomarkers Prev. 2012 Nov;21(11):2108-17. doi: 10.1158/1055-9965.EPI-12-0740. Epub 2012 Oct 30. PMID 23112268